CLINICAL TRIAL: NCT02581904
Title: Evaluation of Closed Incision Negative Pressure Device (Prevena) to Prevent Vascular Wound Complications
Brief Title: Prevena Vascular Groin Wound Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7179
Record Dates: First submitted 2015-10-08; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Wound Infection; Peripheral Arterial Disease; Aneurysm; Surgical Wound Dehiscence
MeSH Terms: conditions — Wound Infection; Peripheral Arterial Disease; Aneurysm; Surgical Wound Dehiscence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Risk - Prevena Care (Experimental): The Prevena device is a product from KCI and is a sterile sponge that covers the closed incision. The device is placed sterile in the operating room and suction is then applied to the sponge for 5-7 days.
  Interventions: Device: Prevena Care
- High Risk - Dry Gauze Dressing Care (Active Comparator): Initial dry gauze dressing will be placed sterile in the operating room and will be changed daily
  Interventions: Device: Dry gauze dressing care
- Low Risk - Dry Gauze Dressing Care (Active Comparator): Initial dry gauze dressing will be placed sterile in the operating room and will be changed daily
  Interventions: Device: Dry gauze dressing care

INTERVENTIONS:
Device: Prevena Care — The Prevena device is a product from KCI and is a sterile sponge that covers the closed incision. The device is placed sterile in the operating room and suction is then applied to the sponge for 5-7 days.
  Other Names: Closed Incision Negative Pressure Device
  Arms: High Risk - Prevena Care
Device: Dry gauze dressing care — Initial dry gauze dressing will be placed sterile in the operating room and will be changed daily
  Arms: High Risk - Dry Gauze Dressing Care; Low Risk - Dry Gauze Dressing Care

SUMMARY:
The purpose of this study is to determine if the application of a negative pressure dressing intraoperatively (Prevena; KCI, Inc) to vascular groin incisions decreases the wound complication rate in high risk patients.

DETAILED DESCRIPTION:
The study randomizes patients (1:1) considered high risk, according to a specific set of risk factors, for wound complications into standard post-op dressings vs. Prevena vacuum dressing. The wounds will then be assessed for wound complications in the 30 days postoperatively. Wound complications include breakdown, infection and lymph leak. Patients not considered high risk will have standard post-op dressings and followed similarly to controls. The investigators will also assess economic impact of negative pressure dressing on length of stay and overall inpatient costs.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a femoral incision during vascular reconstruction or repair will be considered for study

Exclusion Criteria:

* Emergency procedure
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Groin Wound Complication | 30 days
  Composite measure including wound dehiscence (skin or fascia), lymph leak (seroma or fistula), infection (deep or superficial), or hematoma

SECONDARY OUTCOMES:
Hospital Length of stay | 30 days
Return to Operating Room | 30 days
Hospital Readmission | 30 days
  Readmission for wound complication
Index Hospital Cost | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul DiMuzio, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- [Derived] Cristino MA, Nakano LC, Vasconcelos V, Correia RM, Flumignan RL. Prevention of infection in aortic or aortoiliac peripheral arterial reconstruction. Cochrane Database Syst Rev. 2025 Apr 22;4(4):CD015192. doi: 10.1002/14651858.CD015192.pub2. PMID 40260835
- [Derived] Kwon J, Staley C, McCullough M, Goss S, Arosemena M, Abai B, Salvatore D, Reiter D, DiMuzio P. A randomized clinical trial evaluating negative pressure therapy to decrease vascular groin incision complications. J Vasc Surg. 2018 Dec;68(6):1744-1752. doi: 10.1016/j.jvs.2018.05.224. Epub 2018 Aug 17. PMID 30126781